CLINICAL TRIAL: NCT01459796
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Long-Term Rilonacept Treatment for the Prevention of Gout Flares
Brief Title: Study of the Safety and Efficacy of Long-Term Rilonacept Treatment for the Prevention of Gout Flares
Acronym: UPSURGE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IL1T-GA-1101
Record Dates: First submitted 2011-10-12; First posted 2011-10-26 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — rilonacept; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection once a week (qw) from Week 1 to Week 51.
  Interventions: Drug: Placebo; Drug: Allopurinol
- Rilonacept 80 mg (Experimental): Two subcutaneous injections of Rilonacept 80 mg (for a total of 160 mg) as a loading dose on Day 1, followed by a single 80 mg injection of Rilonacept qw from Week 1 to Week 51.
  Interventions: Drug: Rilonacept; Drug: Allopurinol

INTERVENTIONS:
Drug: Rilonacept — Rilonacept 160 mg loading dose followed by Rilonacept 80 mg/2 mL injections qw for 52 weeks.
  Arms: Rilonacept 80 mg
Drug: Placebo — Placebo loading dose followed by placebo injections (2 mL) qw for 52 weeks.
  Arms: Placebo
Drug: Allopurinol — Allopurinol 50 or 100 mg, orally daily for 52 weeks as background treatment.

SUMMARY:
The purpose of this study was to determine the safety and tolerability of rilonacept for participants with gout who were initiating allopurinol.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion criteria:

* Male or female participants aged 18 to 80 years;
* Previously met the preliminary criteria of the ARA for the classification of the acute arthritis of primary gout;
* Serum uric acid greater than or equal to 7.5 mg/dL at the screening visit;
* A self-reported history of at least 2 gout flares in the year prior to screening.

Exclusion Criteria:

Key Exclusion criteria:

* Pregnant or nursing, or planning to become pregnant or father a child within 3 months after receiving the last dose of study drug;
* Participants requiring dialysis;
* Participants who had had an organ transplant;
* Persistent chronic or active infections;
* Previous exposure to rilonacept;
* Use of allopurinol, benzbromarone, febuxostat, probenecid or sulfinpyrazone within 84 days prior to the screening visit.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (74):
- United States (74):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Searcy, Arkansas
  - Concord, California
  - La Jolla, California
  - Long Beach, California
  - Whittier, California
  - Denver, Colorado
  - Trumbull, Connecticut
  - Washington D.C., District of Columbia
  - Clearwater, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Venice, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Meridian, Idaho
  - Avon, Indiana
  - Brownsburg, Indiana
  - Evansville, Indiana
  - Bowling Green, Kentucky
  - Elizabethtown, Kentucky
  - Owensboro, Kentucky
  - New Orleans, Louisiana
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Fall River, Massachusetts
  - Edina, Minnesota
  - St Louis, Missouri
  - Kalispell, Montana
  - Omaha, Nebraska
  - Brooklyn, New York
  - Cary, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Carlisle, Ohio
  - Portland, Oregon
  - Huntingdon Valley, Pennsylvania
  - Johnstown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Rock Hill, South Carolina
  - Simpsonville, South Carolina
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 60 study sites in the United States (US) from 12 November 2011 to 02 November 2012. A total of 485 participants were screened in the study.
Pre-assignment Details: Out of 485 participants, 220 were randomized and treated in the study. Participants were randomized in 4:3 ratio to receive either Rilonacept 80 mg or Placebo.
Period: Overall Study
Arm/Group | Placebo | Rilonacept 80 mg
Started | 94 | 126
Completed | 0 | 0
Not Completed | 94 | 126
Not completed — Non compliance with protocol | 2 | 4
Not completed — Adverse Event | 5 | 5
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lost to Follow-up | 5 | 4
Not completed — Reason unspecified | 1 | 2
Not completed — Decision by the sponsor | 75 | 108

BASELINE CHARACTERISTICS:
Population: Baseline population included full analysis set (FAS) comprising of all randomized participants who received any study medication and was based on treatment allocated by Interactive web response system (IWRS) at randomization (as randomized).
Groups:
- Placebo: Two subcutaneous injections of Placebo (for Rilonacept) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 51.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilonacept 80 mg | Total
Number analyzed (Participants) | 94 | 126 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.69) | 52.1 (11.18) | 51.9 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 86 | 111 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 87 | 120 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 9 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 16 | 27 | 43
  White | 75 | 87 | 162
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (time from the administration of first dose of study drug up to and including 35 days after the last dose of study drug). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Day 1 to Day 392 (Week 56)
Population: Safety analysis set (SAF) that included all randomized participants who received any study medication and was based on the treatment received (as treated).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 80 mg
Number analyzed (Participants) | 94 | 126
percentage of participants
  With at least one TEAE | 68.1 | 68.3
  With TEAEs related to study drug | 12.8 | 19.0
  With serious TEAEs | 5.3 | 4.0
  With TEAEs resulting in study drug discontinuation | 10.6 | 6.3
  With TEAEs resulting in death | 0.0 | 0.0

2. Secondary Outcome: Percentage of Participants With at Least One Gout Flare From Day 1 to Day 168 (Week 24)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain; and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least one gout flare at Week 24 was to be reported for this outcome measure.
Time Frame: Day 1 to Day 168 (Week 24)
Population: As per sponsor's discretion, the study was discontinued due to which data for this outcome measure was not collected and hence, not analyzed and reported.
Arm/Group | Placebo | Rilonacept 80 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With at Least Two Gout Flares From Day 1 to Day 168 (Week 24)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least two gout flares at Week 24 was to be reported for this outcome measure.
Time Frame: Day 1 to Day 168 (Week 24)
Population: as for outcome 2
Arm/Group | Placebo | Rilonacept 80 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With at Least One Gout Flare From Day 1 to Day 364 (Week 52)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain; and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least one gout flare at Week 52 was to be reported for this outcome measure.
Time Frame: Day 1 to Day 364 (Week 52)
Population: as for outcome 2
Arm/Group | Placebo | Rilonacept 80 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With at Least Two Gout Flares From Day 1 to Day 364 (Week 52)
Description: Gout flare was defined as acute articular pain typical of a gout attack that required treatment with an anti-inflammatory therapeutic: had at least 3 of the following 4 signs or symptoms: joint swelling, tenderness, redness, and pain, and with at least 1 of the following: rapid onset of pain, decreased range of motion, joint warmth or other symptoms similar to a prior gout flare. Percentage of participants with at least two gout flares at Week 52 was to be reported for this outcome measure.
Time Frame: Day 1 to Day 364 (Week 52)
Population: as for outcome 2
Arm/Group | Placebo | Rilonacept 80 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Rescue Medication From Day 1 to Day 364 (Week 52)
Description: Participants who required rescue medication after having 2 or more gout flares during the treatment period were evaluated.
Time Frame: Day 1 to Day 364 (Week 52)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rilonacept 80 mg
Number analyzed (Participants) | 94 | 126
percentage of participants | 22.3 | 8.7

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 56) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the administration of first dose of study drug up to and including 35 days after the last dose of study drug). Analysis was performed on safety analysis set (SAF).
Arm/Group | Placebo | Rilonacept 80 mg
Serious Adverse Events (participants affected / at risk) | 5/94 | 5/126
Other Adverse Events (participants affected / at risk) | 31/94 | 43/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Rilonacept 80 mg (N=126)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2)
Drug interaction (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Rilonacept 80 mg (N=126)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 9 (9)
Nausea (Gastrointestinal disorders) | 5 (23) | 2 (2)
Injection site erythema (General disorders) | 2 (3) | 9 (27)
Nasopharyngitis (Infections and infestations) | 3 (3) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (9)
Headache (Nervous system disorders) | 6 (11) | 11 (55)
Hypertension (Vascular disorders) | 2 (5) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI/Institution will provide a copy of any publication to Sponsor prior to submission for review. Sponsor may request to remove confidential information from submission, provided that removal does not preclude the complete and accurate presentation and interpretation of the study results.